CLINICAL TRIAL: NCT03645603
Title: Efficacy and Safety of Dexmedetomidine During Weaning From Analgesia and Sedation in Pediatric Intensive Care Unit. A Multicenter, Double-blind, Randomized Controlled Trial.
Brief Title: Efficacy and Safety of Dexmedetomidine During Weaning From Analgesia and Sedation in PICU (TIP-15-01)
Acronym: TIP-15-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: futility reasons
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Azienda Ospedaliera di Padova (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Maria Cristina Mondardini, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT 2015-002114-80 OsSC
Record Dates: First submitted 2018-08-17; First posted 2018-08-24 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Withdrawal Syndrome
Keywords: pediatrics; dexmedetomidine; analgesia; sedation; pediatric intensive care unit; abstinence syndrome; assessment tool
MeSH Terms: conditions — Substance Withdrawal Syndrome; Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine 100 mcg/ml concentrate solution. Continuous iv infusion. Start dose 0.4 mcg/kg/h, increases by 0.2 mcg/kg/h until 0.8 mcg/kg/h (half dose for neonates). If withdrawal symptoms appear the dose can be increased to a maximum of 1.4 mcg/Kg/h.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): saline solution for IV infusion. The administration of infusion will follow the experimental drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — intravenous infusion
  Other Names: Dexdor, Precedex
  Arms: Dexmedetomidine
Drug: Placebo — intravenous infusion of physiological saline solution to mimic dexmedetomidine infusion
  Other Names: physiological saline solution
  Arms: Placebo

SUMMARY:
This interventional study evaluates the efficacy of dexmedetomidine during weaning from analgesic and sedative drugs in reducing the occurrence of the withdrawal syndrome in PICU. All enrolled patients will undergo the same weaning regimen one half will receive dexmedetomidine while the other will receive a placebo.

DETAILED DESCRIPTION:
Children admitted to PICU need of analgesic and sedative drugs. Prolonged treatment can lead to undesirable effects as dependence and tolerance. Patients that have developed dependence may develop the withdrawal syndrome (WS) during the analgesics and sedatives weaning process.

Withdrawal symptoms are due to central nervous system excitement, gastrointestinal disturbance, and sympathetic system activation. The incidence of withdrawal syndrome is variable between 17 and 57% a recent study reported an incidence of 64.6% of WS in Italian PICUs. The prevention strategies are addressed to the restriction of drug exposure and to the gradual tapering of infusion. However, these strategies have weak evidence of effectiveness. In this study, the investigators hypothesize that dexmedetomidine may be useful and effective during the weaning of analgosedation drugs in PICU, in preventing the withdrawal syndrome. The primary aim of the study is to evaluate the efficacy of dexmedetomidine in reducing the occurrence of the WS. Secondary aims are to evaluate the dexmedetomidine safety during the weaning, the effective dose range, and the efficacy in reducing the duration of the weaning, of the mechanical ventilation, and of the length of PICU stay. Efficacy will be compared among pediatric age groups, gender, race, Pediatric Index of Mortality (PIM3) score, and length of the analgosedation treatment.

Patients admitted to the PICU that meets the inclusion criteria, will be randomly assigned to one of the two treatment groups: treatment A (dexmedetomidine) or treatment B (placebo).

Twenty-four hours before the start of the weaning an intravenous infusion of dexmedetomidine/placebo will start. After 24 hours of dexmedetomidine infusion, the weaning regimen will begin following the subsequent indications: 10% reduction of the dose every 12 hours. The withdrawal assessment tool version 1 (WAT-1) is the selected scale to evaluate the occurrence of the WS. Patients with a score of WAT-1 <3 continue the weaning regimen. Patients with a score ≥3 increase the dose of dexmedetomidine/placebo until the next WAT-1 score control and temporarily stop the planned 10% dose reduction. If the next WAT-1 score decreased by at least 1 point from the previous score, the weaning program restarted (10% reduction) without further changes in the dose of dexmedetomidine/placebo until the subsequent score. The 'acute withdrawal crisis' will be treated with a rescue dose of the opioid and/or benzodiazepine in use repeatable until resolution of the crisis. Once analgesics and sedatives weaning is complete, dexmedetomidine will gradually discontinue. Five days after discharge from PICU, a follow-up visit will be performed.

The sample size estimate is 80 participants for each of the two groups for a total of 160 patients recruited within a period of two years.

ELIGIBILITY:
Inclusion Criteria:

* Continuous analgesic and sedative endovenous treatment for at least 5 days
* Invasive or non-invasive mechanical ventilation
* Clinical conditions that allow by clinical judgment the start of analgosedation weaning
* Post-natal age ≥ 7 days and PMA beyond the 37 weeks
* Written informed consent obtained

Exclusion Criteria:

* Hemodynamic instability
* Cardiac bundle-branch block of 2 or 3 degree
* Hypersensitivity to the alpha-agonists
* Persistent fever of unknown origin or sensitivity to malignant hyperthermia
* Use of alpha-agonist (clonidine or dexmedetomidine) in the last 30 days

Ages: 7 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Change in Withdrawal Assessment Tool (WAT-1) scale | time 0 start dexmedetomidine and every 12 hours post-start dexmedetomidine for 7 days
  WAT-1 score recorded every 12 hours.The score ranges from 0 to 12, a score ≥3 indicates the presence of signs/symptoms of withdrawal.

SECONDARY OUTCOMES:
Change in heart rate | 0,1, 2, 12, 24 hours post-start dexmedetomidine and then every 12 hours for 7 days
  changes in heart rate will be recorded when their value differs more than 20% by the patient's baseline values.
Change in Systolic Blood Pressure | 0,1, 2, 12, 24 hours post-start dexmedetomidine and then every 12 hours for 7 days
  changes in Systolic Blood Pressure will be recorded when their value differs more than 20% by the patient's baseline values.
Change in Diastolic Blood Pressure | 0,1, 2, 12, 24 hours post-start dexmedetomidine and then every 12 hours for 7 days
  changes in Diastolic Blood Pressure will be recorded when their value differs more than 20% by the patient's baseline values.

OTHER OUTCOMES:
Change in Opioid dose | 7 days
  verification of adherence to weaning regimen
Change in Sedative dose | 7 days
  verification of adherence to weaning regimen

CONTACTS AND LOCATIONS:
Overall Officials: Maria C. Mondardini, MD, Study Chair — Azienda Ospedaliero Universitaria di Bologna Policlinico S.Orsola-Malpighi
Locations (1):
- PICU Policlinico S.Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amigoni A, Mondardini MC, Vittadello I, Zaglia F, Rossetti E, Vitale F, Ferrario S, Savron F, Coffaro G, Brugnaro L, Amato R, Wolfler A, Franck LS; Network of Paediatric Intensive Care Unit Study Group (TIPNet). Withdrawal Assessment Tool-1 Monitoring in PICU: A Multicenter Study on Iatrogenic Withdrawal Syndrome. Pediatr Crit Care Med. 2017 Feb;18(2):e86-e91. doi: 10.1097/PCC.0000000000001054. PMID 28157809
- [Derived] Mondardini MC, Daverio M, Caramelli F, Conti G, Zaggia C, Lazzarini R, Muscheri L, Azzolina D, Gregori D, Sperotto F, Amigoni A. Dexmedetomidine for prevention of opioid/benzodiazepine withdrawal syndrome in pediatric intensive care unit: Interim analysis of a randomized controlled trial. Pharmacotherapy. 2022 Feb;42(2):145-153. doi: 10.1002/phar.2654. Epub 2021 Dec 21. PMID 34882826
- [Derived] Mondardini MC, Sperotto F, Daverio M, Caramelli F, Gregori D, Caligiuri MF, Vitale F, Cecini MT, Piastra M, Mancino A, Pettenazzo A, Conti G, Amigoni A. Efficacy and safety of dexmedetomidine for prevention of withdrawal syndrome in the pediatric intensive care unit: protocol for an adaptive, multicenter, randomized, double-blind, placebo-controlled, non-profit clinical trial. Trials. 2019 Dec 11;20(1):710. doi: 10.1186/s13063-019-3793-6. PMID 31829274

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT03645603/Prot_SAP_000.pdf